CLINICAL TRIAL: NCT01323738
Title: Effect of Psychoeducation on Motivation to Change in Traumatized Alcoholics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Konstanz (Other)
Responsible Party: Dr. Michael Odenwald, University of Konstanz
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: UKonstanzMOdenwald2009-1
Record Dates: First submitted 2009-12-22; First posted 2011-03-28 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Alcoholic Intoxication, Chronic
Keywords: Psychoeducation; Group Control
MeSH Terms: conditions — Alcoholism | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment as Ususal (No Intervention): Patients participate in the Treatment as Usual including a non-specific information group.
- Psychoeducation (Experimental): Intervention group
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — Psychoeducation group on stress and how it relates to alcohol use, 4 sessions a 45 minutes
  Other Names: The manualized group intervention we developed for this study recently was named TARGET,; which reads as "Trauma- and Alcohol-Related Group Education and motivation Therapy"
  Arms: Psychoeducation

SUMMARY:
Many people suffering from alcohol dependence have a history of exposure to stressful life situations, such as childhood physical or emotional misuse. Often, there's a functional relationship between drinking and emotional problems related to past traumatic experiences, i.e. drinking to forget. However, alcohol treatment often does not include interventions to support patients to cope better with past life experiences. On the other hand, most alcoholics are poorly motivated to participate in long-term rehabilitative treatments after detoxification. In the proposed study, the investigators will study the effects of a brief psycho-educational group intervention during detoxification treatment on motivation to change and the willingness to accept further treatment.

The investigators will use a group comparison design (intervention versus "TAS" control group). In month 1, patients take part in Treatment as Usual (TAS), including a unspecific information group. In month 2, the information group is replaced by the psychoeducational group (intervention). Ward staff selects patients for the groups, irrespective of intervention or TAS. Selection criteria are: absence of severe withdrawal and cognitive impairment. Absence of severe co-morbid psychiatric disorder (e.g. schizophrenia or suicidal crisis). The group sessions will take place in groups of up to 15 patients and will include 4 structured sessions (45 min each). Main content if the intervention group is to highlight and discuss the association between stress, Posttraumatic Stress Disorder and drinking. Patients will also be informed about the different treatment options available in the region.

At entry, patients are asked to fill in the German versions of the University of Rhode Island Change Assessment (URICA; McConnaughy, Prochaska, & Velicer, 1983; German: Heidenreich, Hoyer & Fecht; 2001) and the Trauma History Questionnaire (THQ; Green, 1996; German: Maercker, 2002). At discharge, patients are asked to fill in the URICA.

The investigators expect that specific information on the association between stress and drinking will increase the patients' motivation to participate in further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol Dependence
* Regular admission to detoxification unit

Exclusion Criteria:

* Severe withdrawal
* Severe cognitive impairment
* Severe comorbid psychiatric conditions (schizophrenia, suicidal crisis)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
University of Rhode Island Change Assessment (URICA) | Pre and Post (day 1, day 15 (average))
  Pre-assessment is at entry in in-patient alcohol detoxification treatment, post-assessment is at day of discharge. On average, the two measurements are 15 days apart.
Detoxification treatment completion | 15 days (average treatment duration)
  It was evaluated how many subjects in both treatment arms and among traumatized and non-traumatized in each arm ended the detoxification treatment prematurely, i.e. discharge against medical advice or disciplinary discharge.
number of days in detoxification treatment | 15 days (average treatment duration)
  The number of days in detoxification treatment is a simple count of days of treatment between day of detoxification treatment entry and day of discharge

SECONDARY OUTCOMES:
adverse events | between admission and discharge
  Adverse events were assessed during the detoxification treatment for patients taking part in the information group (TAU) or TARGET group (intervention), i.e. suicide attempts, psychiatric decompensation, aggressive behaviors, relapse of alcohol use. These events were recorded by the social worker who participated routinely in the three daily team meetings during which the situation of each patient was briefly discussed.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Odenwald, PhD, Principal Investigator — University of Konstanz
Locations (1):
- Center for Psychiatry Reichenau, Reichenau, Germany